CLINICAL TRIAL: NCT03428295
Title: Assessments of Hybrid Closed Loop and Fully Automated Closed Loop Dose Safety Artificial Pancreas Device in Type 1 Diabetes in a Hospital Clinical Research Setting
Brief Title: Dose Safety Hybrid Closed Loop and Fully Automated Closed Loop Artificial Pancreas Device in CRC
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Further software development is required.
Sponsor: Dose Safety Inc. (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Benaroya Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APS4; 2R44DK104317-03 (NIH)
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Glucose, Low Blood; Glucose, High Blood
Keywords: artificial pancreas; automated insulin delivery; hybrid closed loop; APDS; fully automated closed loop

STUDY DESIGN:
Intervention Model Description: Experimental: Single Cohort in CRC This study is a single-arm, multi-center, observational clinical trial being conducted in a Clinical Research Center (CRC) setting. Intervention: Device: Dose Safety Artificial Pancreas (AP) System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental: Single Cohort in CRC (Experimental): This study is a single-arm, single-center, observational clinical trial being conducted in a Clinical Research Center (CRC) setting.
  Interventions: Device: Dose Safety AP system

INTERVENTIONS:
Device: Dose Safety AP system — Device will be used to automatically dose insulin

SUMMARY:
The objective of this study is to test two different operating modes of the latest version of the Dose Safety artificial pancreas system (APS), the Dose Safety Controller (DSC version 2.3), in a population of subjects with type 1 diabetes (TID) in a hospital CRC setting. The first mode is the Fully Automated Closed Loop (FACL) mode, in which all insulin delivery is directed by the controller and the second mode is the Hybrid Closed Loop (HCL) mode, in which insulin delivery is a hybrid between controller directed delivery and user directed insulin delivery. There will be two study arms: HCL and FACL. No comparisons will be made between the two arms.

DETAILED DESCRIPTION:
3.1 Overview Two independent questions will be addressed in this study. For evaluation of the safety and efficacy of the hybrid closed loop (HCL), participants will use the hybrid closed loop during and after a standardized meal on the clinical research center. For evaluation of the safety and efficacy of the fully automated closed loop (FACL), participants will use the system for a 24 hour clinical research center stay incorporating meals and standardized exercise. Safety and efficacy will be evaluated by descriptive outcomes including number of completed studies and glycemic control.

3.2 Eligibility. Participants will be recruited from the Diabetes Registry at the Benaroya Research Institute. Eligibile participants may enroll in the HCL, the FACL, or both studies.

HCL Study visit, Day 1 (~7 hours total): The below times are approximate and may be adjusted to accommodate the CRC schedule. Prior to arrival at the CRC, participants will be asked to eat their normal breakfast and take their usual amount of insulin based on BG and carbohydrate content before 8am. Once at the CRC, participants will be able to drink water ad lib, but no food other than the prescribed meals can be eaten, unless hypoglycemia intervention is necessary. Participants will be required to check FSBG before the meal and calibrate if the FSBG value varies by >30% from CGM value.

FACL Study visit, Day 1 (~ 23 hours total): The below times are approximate and may be adjusted to accommodate the CRC schedule. Prior to arrival at the CRC, participants will be asked to eat their normal breakfast and take their usual amount of insulin based on BG and carbohydrate content before 8 am. Once arrived at the CRC, participants will be able to drink water, but no food other than the prescribed meals can be eaten, unless hypoglycemia intervention is necessary. Participants will be required to check FSBG before meals, at bedtime and at 0300. They will calibrate if the FSBG value varies by >30% from the CGM value. They will calibrate the CGM every 12 hours as recommended by Dexcom.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have type 1 diabetes for greater than 1 year
* Have a hemoglobin A1c less than 9.0%
* Participants in the FACL arm must report that they engage in aerobic exercise at least 30 minutes three times weekly
* If participants in the FACL arm are age >35 OR duration of T1D >15 years OR history of T1D complications (proliferative retinopathy, nephropathy, peripheral vascular disease, autonomic neuropathy), participant must have EKG within normal limits obtained within last 6 months of study date
* Age 18-70
* Fluent and literate in English
* Use of an insulin pump for ≥ 3 months
* Use of a CGM/sensor for ≥ 5 days/week for ≥3 months
* Must have a diabetes care provider
* Use of an effective birth control method for women who are sexually active and of childbearing potential
* Willing and able to give informed consent

Exclusion Criteria:

* History of ≥ 1 episode of severe hypoglycemia (defined as hypoglycemia leading to loss of consciousness, seizure, or requiring assistance) in the previous 6 months
* History of ≥ 1 episode of DKA in the previous 6 months
* History of cardiovascular disease, characterized by any of the following:

  * Prolonged QT or arrhythmia
  * History of myocardial infarction within the past 6 months
  * History of ischemia on functional cardiac exam within the last year
  * History of left ventricular ejection fraction < 30%
* Uncontrolled hypertension (SBP > 160 mmHg or DBP > 100 mmHg)
* Current use of a beta blocker
* Stage 3 or greater renal disease
* Untreated thyroid disease
* History of substance abuse
* Current or previous use of medications for control of a seizure disorder
* Enrolled in another clinical trial in which they received investigational drug in the last 12 weeks
* Inability to comply with protocol
* Pregnant or breast feeding
* Use of medications other than insulin to control glucose
* Chronic corticosteroid use
* Pre-existing medical conditions deemed by study investigator to interfere with the study or increase risks of study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of time in hypoglycemic range | 36 hours
  defined as <70 mg/dL
Percentage of time in severe hyperglycemic range | 36 hours
  defined as >/=250 mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Dose Safety, Redmond, Washington, United States

IPD SHARING:
Plan to Share IPD: No